CLINICAL TRIAL: NCT03711058
Title: A Phase I/II Study of PI3Kinase Inhibition (Copanlisib) and Anti-PD-1 Antibody Nivolumab in Relapsed/Refractory Solid Tumors With Expansions in Mismatch-repair Proficient (MSS) Colorectal Cancer
Brief Title: Study of PI3Kinase Inhibition (Copanlisib) and Anti-PD-1 Antibody Nivolumab in Relapsed/Refractory Solid Tumors With Expansions in Mismatch-repair Proficient (MSS) Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bayer (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J1887; IRB00175864 (Other: JHM IRB); CA209-8LC (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Unresectable or Metastatic Microsatellite Stable (MSS) Solid Tumor; Microsatellite Stable (MSS) Colon Cancer
Keywords: Immunotherapy; Nivolumab; Copanlisib; Unresectable; Metastatic; PD-1; P13K; Antibody; Solid Tumors; Colon Cancer; MSS; Mismatch-repair proficient; Microsatellite stable
MeSH Terms: conditions — Spinocerebellar Degenerations; Colonic Neoplasms; Neoplasm Metastasis | interventions — copanlisib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I - Copanlisib and Nivolumab (De-Escalation) (Experimental)
  Interventions: Drug: Copanlisib; Drug: Nivolumab
- Phase II /Arm A-P13K mutation/Copanlisib and Nivolumab (Experimental)
  Interventions: Drug: Copanlisib; Drug: Nivolumab
- Phase II/Arm B -P13K wild type /Copanlisib and Nivolumab (Experimental)
  Interventions: Drug: Copanlisib; Drug: Nivolumab

INTERVENTIONS:
Drug: Copanlisib — Copanlisib will be administered as a 60 minute IV infusion (-5min/+10min) at a dose of 45 mg - 60 mg IV. Copanlisib will be administered once a week (days 1, 8, and 15 or Day 1 and Day 15 of each 28 day cycle).
  Drug: 45 or 60 mg IV
  Other Names: Bay 80-6946
Drug: Nivolumab — Nivolumab 480 mg will be administered as a 30 minute IV infusion (-5min/+10min) on Day 1 of each 28 day cycle.
  Drug: 480 mg IV
  Other Names: OPDIVO, Bay 80-6946

SUMMARY:
A phase I/II study of PI3Kinase inhibition (copanlisib) and anti-PD-1 antibody nivolumab in relapsed/refractory solid tumors with expansions in mismatch-repair proficient (MSS) colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Ability to understand and willingness to sign a written informed consent document.
* Phase I: Must have received all curative treatment options and at least 2 lines of systemic therapy.
* Phase II: Must have received at least 2 lines of systemic therapy including a fluoropyrimidine, oxaliplatin, and irinotecan-containing regimen. KRAS/NRAS/BRAF wildtype patients must have received or refused anti-EGR.
* Must have received all curative treatment options and at least 2 lines of systemic and standard therapy.
* Must have measurable disease based on RECIST 1.1
* Must have biopsiable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy of greater than 3 months.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests within 21 days of initial study drug.
* Men must use acceptable form of birth control while on study.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.

Exclusion Criteria:

* Prior treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti- PD-L2, anti-CTLA4, etc.).
* Prior therapy with a PI3K inhibitor
* Chemotherapy, target small molecule therapy, investigational therapy, or surgery within 4 weeks prior to first dose of treatment.
* Has received prior radiotherapy within 2 weeks prior to the start of treatment.
* Patient who is receiving or have received any other investigational agents within 4 weeks prior to the first dose of treatment.
* Has received a live vaccine 30 days prior to the first dose of study drug.
* Has known additional malignancy that is progressing or requires active treatment..
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has symptomatic ascites or has required a paracentesis in the last 12 weeks.
* Hypersensitivity reaction to study drug.
* Patients diagnosed of immunodeficiency or are on any immunosuppressive agents within 7 days prior to first dose of study drug.
* Has active autoimmune disease that has required systemic treatment in the past 12 months, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Infection with HIV or hepatitis B or C.
* Cytomegalovirus polymerase chain reaction (CMV PCR) positive.
* Known history or concurrent interstitial lung disease.
* Type I diabetes or Type II diabetes requiring treatment with a sulfonylurea, meglitinide, or insulin at screening.
* Uncontrolled cardiovascular disease.
* Patient with uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Use of anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Use of CYP3A4 inhibitors and inducers within 2 weeks of starting study drug and throughout treatment.
* Any arterial or venous thrombotic or embolic events within 3 months of start of study drug.
* Non-healing wound, ulcer, or fracture.
* Patients with evidence or history of bleeding condition.
* Had a blood or platelet transfusion within 7 days of Cycle 1 Day 1 treatment.
* Seizure disorder requiring anti-seizure medication.
* Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures.
* Are pregnant or breastfeeding.
* Unwilling or unable to follow the study schedule for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Morschhauser F, Machiels JP, Salles G, Rottey S, Rule SAJ, Cunningham D, Peyrade F, Fruchart C, Arkenau HT, Genvresse I, Liu L, Kochert K, Shen K, Kneip C, Pena CE, Grevel J, Zhang J, Cisternas G, Reschke S, Granvil C, Awada A. On-Target Pharmacodynamic Activity of the PI3K Inhibitor Copanlisib in Paired Biopsies from Patients with Malignant Lymphoma and Advanced Solid Tumors. Mol Cancer Ther. 2020 Feb;19(2):468-478. doi: 10.1158/1535-7163.MCT-19-0466. Epub 2019 Oct 16. PMID 31619463

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants (1 from Phase 1, 4 from Phase 2 Cohort A and 4 from Phase 2 Cohort B) were excluded from analysis because they did not receive the study drug.
Groups:
- Phase I - Dose Finding: Copanlisib will be administered as a 60-minute IV infusion (-5min/+10min) at one of three dose levels:
  Dose Level 1: 60mg on Day 1, 8, and 15
  Dose Level -1: 60mg on Day 1 and 15
  Dose Level -2: 45 mg on Day 1 and 15
  Nivolumab 480 mg will be administered as a 30-minute IV infusion (-5min/+10min) on Day 1 of each cycle.
  Cycle length is 28 days.
  Only Dose Level 1 was tested.
- Phase II /Cohort A - PI3K Mutation; Phase II /Cohort B - PI3K Wild Type: Copanlisib 60 mg will be administered as a 60-minute IV infusion (-5min/+10min) on Day 1, 8, and 15 of each 28-day cycle.
  Nivolumab 480 mg will be administered as a 30-minute IV infusion (-5min/+10min) on Day 1 of each 28-day cycle.
Period: Overall Study
Arm/Group | Phase I - Dose Finding | Phase II /Cohort A - PI3K Mutation | Phase II /Cohort B - PI3K Wild Type
Started (started = enrolled and received at least one dose of study drug) | 6 | 21 | 12
Completed | 6 | 21 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I - Dose Finding: Copanlisib: Copanlisib will be administered as a 60 minute IV infusion (-5min/+10min) at one of three dose levels:
  Dose Level 1: 60mg on Day 1, 8, and 15
  Dose Level -1: 60mg on Day 1 and 15
  Dose Level -2: 45 mg on Day 1 and 15
  Nivolumab: Nivolumab 480 mg will be administered as a 30 minute IV infusion (-5min/+10min) on Day 1 of each cycle.
  Cycle length is 28 days.
  Only Dose Level 1 was tested.
- Phase II/Cohort B - PI3K Wild Type: Copanlisib 60 mg will be administered as a 60-minute IV infusion (-5min/+10min) on Day 1, 8, and 15 of each 28-day cycle.
  Nivolumab 480 mg will be administered as a 30-minute IV infusion (-5min/+10min) on Day 1 of each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Finding | Phase II /Cohort A - PI3K Mutation | Phase II/Cohort B - PI3K Wild Type | Total
Number analyzed (Participants) | 6 | 21 | 12 | 39
Age, Continuous [Median (Full Range); unit: years] | 59.5 [51 to 81] | 57 [43 to 83] | 58.5 [40 to 73] | 58 [40 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 15 | 4 | 21
  Male | 4 | 6 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 20 | 11 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 5 | 1 | 6
  White | 5 | 15 | 10 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 21 | 12 | 39
Eastern Cooperative Oncology Group (ECOG) Classification of Participants [Count of Participants; unit: Participants] — Measure description: The ECOG scale measures performance status , which scores ranging from 0-5: 0=fully active , performs without restrictions, 1=can ambulate,but restricted in physical strenuous activity,2=ambulatory and capable of self care , but unable to work , active for >50%of waking hours,3=limited self care, confined to bed or chair for >50%of waking hours,4=completely disabled, totally confined tp bed/chair,5= deceased
  Participants
    ECOG 0 | 3 | 11 | 4 | 18
    ECOG 1 | 3 | 10 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose Limiting Toxicity
Description: Number of participants experiencing a Dose Limiting Toxicity (DLT) in each dose level. DLT is defined as any of the following study drug-related toxicities occurring during the first cycle of study drug on study:
  * Grade 4 anemia
  * Grade ≥ 3 neutropenia lasting ≥ 14 days
  * Grade ≥ 3 febrile neutropenia
  * Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia with clinically significant bleeding
  * Treatment-related ≥ grade 4 AEs, except transient hyperglycemia
  * Grade ≥ 3 Pneumonitis or recurrent Grade 2 pneumonitis
  * Grade ≥ 3 Nephritis
  * Grade ≥ 3 elevated AST or ALT
  * Grade ≥ 2 eye pain or reduction of visual acuity that does not respond to topical therapy, improve to ≤ grade 1 within 2 weeks of topical therapy, or requires systemic therapy
  * Any other Grade ≥ 3 toxicities (with certain exceptions for transient AEs or asymptomatic labs)
Time Frame: 28 days
Population: Per protocol, Dose Limiting Toxicities (DLTs) were only assessed in Phase I subjects in order to determine the Phase II dose of copanlisib. Since no subjects experienced DLTs in Dose Level 1, this was the only dose level tested.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I - Dose Finding (Dose Level 1): Copanlisib will be administered as a 60-minute IV infusion (-5min/+10min) at Dose Level 1: 60mg on Day 1, 8, and 15 of each 28-day cycle.
  Nivolumab 480 mg will be administered as a 30-minute IV infusion (-5min/+10min) on Day 1 of each 28-day cycle.
Arm/Group | Phase I - Dose Finding (Dose Level 1)
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: 6-month Objective Response Rate (ORR) of Patients Treated With Copanlisib and Nivolumab
Description: The proportion of subjects with partial response (PR) or complete response (CR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Per RECIST 1.1, complete response is defined as disappearance of all target lesions, and partial response is defined as at least a 30% decrease in the sum of diameters of target lesions. Lesions are assessed by CT or MRI.
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Groups:
- Phase II /Cohort A- PI3K Mutation; Phase II /Cohort B- PI3K Wild Type: Copanlisib 60 mg will be administered as a 60-minute IV infusion (-5min/+10min) on Day 1, 8, and 15 of each 28-day cycle.
  Nivolumab 480 mg will be administered as a 30-minute IV infusion (-5min/+10min) on Day 1 of each 28-day cycle.
Arm/Group | Phase I - Dose Finding (Dose Level 1) | Phase II /Cohort A- PI3K Mutation | Phase II /Cohort B- PI3K Wild Type
Number analyzed (Participants) | 6 | 21 | 12
Participants | 0 | 2 | 0

3. Secondary Outcome: Disease Control Rate (DCR) Status at 6 Months.
Description: Percentage of participants achieving stable disease (SD) or better (SD + PR + CR).
  Per RECIST 1.1, complete response is defined as disappearance of all target lesions, partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, stable disease occurs when there is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least 20% increase). Lesions are assessed by CT or MRI.
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Finding | Phase II /Cohort A - PI3K Mutation | Phase II /Cohort B - PI3K Wild Type
Number analyzed (Participants) | 6 | 21 | 12
Participants | 0 | 5 | 3

4. Secondary Outcome: Duration of Response (DOR)
Description: Number of months from the first documentation of a partial or complete response by RECIST 1.1 to date of disease progression. Responses may be documented at any time on the study, including patients responding after the 6-month evaluation used for the primary outcome.
Time Frame: 3 years
Population: Only patients who had a partial or complete response by RECIST were evaluable for duration of response.
Measure: Median (Full Range); unit: months
Arm/Group | Phase I - Dose Finding (Dose Level 1) | Phase II /Cohort A- PI3K Mutation | Phase II /Cohort B- PI3K Wild Type
Number analyzed (Participants) | 0 | 3 | 1
months |  | 20.6 [17.0 to 22.8] | 13.1 [13.1 to 13.1]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Number of months from treatment to disease progression (PD)
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I - Dose Finding (Dose Level 1) | Phase II /Cohort A- PI3K Mutation | Phase II /Cohort B- PI3K Wild Type
Number analyzed (Participants) | 6 | 21 | 12
months | 1.64 [1.38 to NA] — Upper bound confidence interval was not estimable due to insufficient number of events | 1.68 [1.64 to NA] — Upper bound confidence interval was not estimable due to insufficient number of events | 1.82 [1.68 to NA] — Upper bound confidence interval was not estimable due to insufficient number of events

6. Secondary Outcome: Overall Survival (OS)
Description: Number of months from the date of first treatment until death or end of follow-up.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I - Dose Finding (Dose Level 1) | Phase II /Cohort A- PI3K Mutation | Phase II /Cohort B- PI3K Wild Type
Number analyzed (Participants) | 6 | 21 | 12
months | 5.61 [2.4 to NA] — Upper bound confidence interval was not estimable due to insufficient number of events | 6.77 [4.21 to 16.04] | 10.26 [4.8 to NA] — Upper bound confidence interval was not estimable due to insufficient number of events

7. Secondary Outcome: Number of Participants Experiencing Study Drug-related Toxicities
Description: Number of participants experiencing study drug-related adverse events Grade 3 or higher as defined by CTCAE v5.0.
Time Frame: 51 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Finding (Dose Level 1) | Phase II /Cohort A- PI3K Mutation | Phase II /Cohort B- PI3K Wild Type
Number analyzed (Participants) | 6 | 21 | 12
Participants | 5 | 16 | 10

ADVERSE EVENTS:
Time Frame: Up to 51 months
Description: Adverse reporting collection was conducted by regular investigator assessment and laboratory measurements
Arm/Group | Phase I - Dose Finding (Dose Level 1) | Phase II /Cohort A - PI3K Mutation | Phase II /Cohort B - PI3K Wild Type
All-Cause Mortality (participants affected / at risk) | 6/6 | 14/21 | 9/12
Serious Adverse Events (participants affected / at risk) | 3/6 | 11/21 | 6/12
Other Adverse Events (participants affected / at risk) | 6/6 | 21/21 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Finding (Dose Level 1) (N=6) | Phase II /Cohort A - PI3K Mutation (N=21) | Phase II /Cohort B - PI3K Wild Type (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Chylous ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Disease progression (General disorders) | 3 (3) | 4 (4) | 3 (3)
Fever (General disorders) | 1 (1) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Oral Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vocal Cord Paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Finding (Dose Level 1) (N=6) | Phase II /Cohort A - PI3K Mutation (N=21) | Phase II /Cohort B - PI3K Wild Type (N=12)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 5 (21) | 3 (22)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Swollen lymph node (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 3 (4) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (6) | 1 (2)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 6 (15) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (5) | 2 (3)
Belching (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 3 (7) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (7) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 8 (19) | 7 (14)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Esophageal varices (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (7) | 0 (0)
Gastrointestinal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral Mucositis (Gastrointestinal disorders) | 1 (1) | 2 (8) | 4 (8)
Nausea (Gastrointestinal disorders) | 4 (5) | 17 (31) | 8 (12)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 11 (15) | 7 (7)
Chills (General disorders) | 3 (3) | 3 (4) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 3 (9) | 4 (6)
Fatigue (General disorders) | 3 (4) | 13 (17) | 4 (5)
Fever (General disorders) | 1 (1) | 2 (3) | 3 (3)
Malaise (General disorders) | 1 (1) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 2 (3)
Pain at biopsy site (General disorders) | 0 (0) | 2 (2) | 2 (3)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (2)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Thrush (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ALT increased (Investigations) | 0 (0) | 4 (10) | 6 (13)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (5) | 5 (7)
AST increased (Investigations) | 0 (0) | 4 (8) | 4 (11)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (6) | 1 (2)
Cholesterol high (Investigations) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 5 (7) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (4) | 2 (5)
Serum amylase increased (Investigations) | 0 (0) | 4 (8) | 1 (1)
TSH increased (Investigations) | 0 (0) | 2 (7) | 2 (17)
Weight loss (Investigations) | 6 (7) | 10 (16) | 5 (13)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 4 (5) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 3 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (7) | 9 (12) | 7 (10)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (6)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (6) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (7) | 1 (5)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (8) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Benign nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (5) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (8) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 5 (6) | 4 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 6 (14) | 2 (4)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 3 (3) | 10 (18) | 5 (11)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (19) | 11 (38) | 7 (23)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (2) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 1 (11) | 1 (12)
Blurred Vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Toe Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Nail Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Groin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT03711058/Prot_SAP_000.pdf